CLINICAL TRIAL: NCT05627505
Title: Diagnostic and Prognostic Value of Lung Microbiota in Early Lung Infection After Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qingyuan Zhan (Other)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Head of Ward 4, Respiratory and Critical Care Medicine, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: 2022-HX-53
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumonia group: Patients in the MICU after lung transplantation were enrolled, and alveolar lavage fluid was obtained within 48 hours of the patient's surgery, divided into aliquots, and subjected to macrogenomic sequencing, routine microbiological testing and cytokine testing. Patients will be divided into pneumonia group if they had a co-infection at the time of sampling.
  Interventions: Diagnostic Test: metagenomic next-generation sequencing
- control group: Patients in the MICU after lung transplantation were enrolled, and alveolar lavage fluid was obtained within 48 hours of the patient's surgery, divided into aliquots, and subjected to macrogenomic sequencing, routine microbiological testing and cytokine testing. Patients will be divided into non-pulmonary infection （control）group if they had no co-infection at the time of sampling.
  Interventions: Diagnostic Test: metagenomic next-generation sequencing

INTERVENTIONS:
Diagnostic Test: metagenomic next-generation sequencing — Collection of bronchoalveolar lavage fluid
  Other Names: next-generation sequencing

SUMMARY:
The present study is a prospective case-control study. Patients were enrolled post lung transplantation and alveolar lavage fluid was obtained within 48 hours of the patient's surgery, divided into aliquots and subjected to macrogenomic sequencing, routine microbiological testing and cytokine testing. Patients were divided into pulmonary infection and non-pulmonary infection groups based on whether they had a co-infection at the time of sampling. Pulmonary infection was used as the primary study endpoint. To describe and compare the characteristics of the lung microbiota in the two groups and to determine whether variation in the lung microbiota could predict the development of lung infection and prognosis in patients in the early post-transplant period.

DETAILED DESCRIPTION:
Lung infection is a common and serious problem in the perioperative period of lung transplantation, and early diagnosis of lung infection is important, while traditional culture methods are time-consuming and have low positivity rates. Pathogenic detection by macro-genomic sequencing (mNGS) may be useful for early and rapid diagnosis of post-operative infections, and the simultaneous detection of lower respiratory tract microbiota may also be useful for early diagnosis of infections. However, the use of lung microbiota in the perioperative period of lung transplantation in the setting of pulmonary infections is still at an exploratory stage. The present study is a prospective case-control study. Patients in the MICU after lung transplantation were enrolled, and alveolar lavage fluid was obtained within 48 hours of the patient's surgery, divided into aliquots, and subjected to macrogenomic sequencing, routine microbiological testing and cytokine testing. Patients were divided into pulmonary infection and non-pulmonary infection groups based on whether they had a co-infection at the time of sampling. Pulmonary infection was used as the primary study endpoint. To describe and compare the characteristics of the lung microbiota in the two groups and to determine whether variation in the lung microbiota could predict the development of lung infection and prognosis in patients in the early post-transplant period. To explore the diagnostic thresholds of common lung pathogens by macrogenomic sequencing in patients with co-infections in the early post-transplant period

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU for lung transplantation; consent for bronchoscopy; informed consent signed by the patient or their representative.

Exclusion Criteria:

* Patients admitted to ICU for other serious illnesses; patients more than 48 hours after lung transplantation; patients predicted to die within 48 hours; participation in other clinical studies; failure to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU after lung transplantation in China-Japan Friendship Hospital
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of lung infection | Within 48 hours after surgery
  Positive etiology, respiratory symptoms, new infiltrative shadow on chest imaging

IPD SHARING:
Plan to Share IPD: No